CLINICAL TRIAL: NCT00815763
Title: Efficacy and Safety of Ginsenoside-Rd for Acute Ischemic Stroke: A Randomized, Double-Blind, Placebo-Controlled, Phase 3, Multicenter Trial
Brief Title: Efficacy and Safety of Ginsenoside-Rd for Acute Ischemic Stroke
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Xijing Hospital (Other)
Responsible Party: the neurology department of Xijing Hospital, Xijing Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: xijing-002
Record Dates: First submitted 2008-12-29; First posted 2008-12-30 (Estimated); Last update posted 2008-12-30 (Estimated); Status verified 2008-12

CONDITIONS: Ischemic Stroke
Keywords: randomized trial; ischemic stroke; Ginsenoside-Rd
MeSH Terms: conditions — Ischemic Stroke | interventions — ginsenoside Rd

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ginsenoside-Rd 20mg (Experimental): infusion of ginsenoside-Rd 20mg once a day and continued for 14 days
  Interventions: Drug: ginsenoside-Rd
- placebo (Placebo Comparator): infusion placebo (group B)once a day and continued for 14 days
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: ginsenoside-Rd — infusion ginsenoside-Rd 20 mg once a day and continued for 14 day
  Arms: ginsenoside-Rd 20mg
Drug: placebo — infusion placebo once a day and continued for 14 day
  Arms: placebo

SUMMARY:
The purpose of this phase 3 study is to validate the efficacy and safety of ginsenoside-Rd for acute ischemic stroke.

DETAILED DESCRIPTION:
A phase Ⅲ randomized, double-blind, placebo-controlled, multicenter study was conducted to examine the efficacy and safety of ginsenoside-Rd in patients with acute ischemic stroke. Stroke patients were randomized equally to receive a 14-day infusion of placebo or ginsenoside-Rd 20mg. Primary end points were NIHSS scores at 15 days. Secondary end points were NIHSS scores and the Barthel index at 8 days, the Barthel index and the modified Rankin scale at 15 days and 90 days. The safety end points included serious and nonserious adverse events, laboratory values and vital signs. Analysis was by intention to treat.

ELIGIBILITY:
Inclusion Criteria:

* between 18 to 75 years
* the first episode
* from onset to admission within 72 hours
* NIHSS scores:5~22

Exclusion Criteria:

* had other intracranial pathologies (e.g., tumor, infection)
* had a neurologic or psychiatric disease
* had a coexisting condition that limited their life expectancy
* had significant drug or alcohol misuse
* had high-grade carotid artery stenosis for which surgery was planned
* were pregnant or nursing
* participated in a clinical trial with an investigational drug or device within the past 3 months
* were unlikely to be available for follow-up

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 390 (Actual)
Dates: Start 2006-09; Primary Completion 2008-06 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
the modified Rankin scale | 90 days

SECONDARY OUTCOMES:
NIHSS scores | 8 days
NIHSS scores | 15 days
the Barthel index | 8 days
the Barthel index | 15 days
the modified Rankin scale | 15 days

CONTACTS AND LOCATIONS:
Overall Officials: Gang Zhao, MD, Study Director — the Department of Neurology , Xijing Hospital; Xuedong Liu, MD, Study Chair — the Department of Neurology, Xijing Hospital
Locations (1):
- the Department of Neurology , Xijing Hospital, Xi'an, Shaanxi, China